CLINICAL TRIAL: NCT01416792
Title: Outcomes & Biochemical Parameters Following Cardiac Surgery: Effects of Transfusion of Residual Blood Using Centrifugation and Multiple-Pass Hemofiltration
Brief Title: Centrifugation vs. Multiple-pass Hemofiltration of the Residual Cardiopulmonary Bypass Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatoon Health Region (Other)
Responsible Party: Principal Investigator, Erick McNair, Clinical Perfusionist, Adjunct Professor, Department of Surgery, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Multiple-pass hemofiltration
Record Dates: First submitted 2011-06-07; First posted 2011-08-15 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2011-09

CONDITIONS: Coronary Artery Disease; Heart Valve Diseases
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases | interventions — Centrifugation; Hemofiltration

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multiple-pass hemofiltration (Experimental)
  Interventions: Procedure: Centrifugation; Procedure: Multiple-pass hemofiltration

INTERVENTIONS:
Procedure: Centrifugation
  Other Names: Cell washing
Procedure: Multiple-pass hemofiltration — The residual volume from the CPB circuit is pumped though a hemofilter for multiple passes removing the crystalloid component thereby concentrating the plasma.
  Other Names: Hemofiltration

SUMMARY:
Traditional cardiac surgery requires patient connection to the Cardiopulmonary Bypass (CPB) apparatus which takes over the function of the heart and lungs while the surgeon performs the necessary surgery. The residual blood left in the CPB equipment (1.5-2.0 L) is centrifuged and washed leaving only red blood cells (RBCs) suspended in a saline solution. The RBCs are reinfused into the patient as needed by the anesthesiologist. The main problem with this technique is that many of the important components of the blood such as plasma proteins and clotting factors are discarded through cell washing. This study will explore a novel method (multiple-pass hemofiltration) of processing the residual pump blood which will allow the patient to receive their own whole blood with minimum waste of important components. The newer method of processing the residual pump volume has also been termed off-line modified ultrafiltration (off-line MUF) and is similar to the process that the kidneys use to filter the blood. It is hypothesized that multiple-pass hemofiltration of the residual CPB volume will reduce the occurrence of inflammatory responses, preserve plasma proteins, and decrease allogenic blood exposure and improve clinical outcomes as compared to centrifugation.

DETAILED DESCRIPTION:
This study is being performed because the traditional method of recovery of the residual volume of blood from the cardiopulmonary bypass circuit involves centrifugation and washing of whole blood with a saline solution. This process is sufficient for the recovery of red blood cells however; it results in the discarding of other important components of the blood. The removal of white blood cells, plasma proteins and clotting factors may result in an increased risk of a adverse outcomes during the post-operative period. The new technique our team wants to investigate returns a greater proportion of the patients' whole blood for reinfusion. Our study objectives are to compare the two techniques and determine which technique produces the safest most reliable method of blood processing to help the patient have a smooth, short, transfusion free post-operative period in the intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* all males and females that will be receiving open heart surgery (Coronary Artery Bypass Grafts and / or Valve repair/replacement) during the study period.

Exclusion Criteria:

* history of bleeding disorders
* history inflammatory diseases rheumatoid arthritis

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | Baseline, Hemodilution and 12-hours post-operatively in ICU
  Serum hemoglobin will be measured from the patient at baseline, after hemodilution, and at 12-hours post-operatively in the ICU.
Albumin | baseline, hemodilution and 12-hours post-operatively in ICU
  Serum albumin in g/L will be measured at baseline, hemodilution and 12-hours post-operatively in ICU.
Total Protein | Baseline, hemodilution, and-12 hours post-operatively in ICU
  Serum total protein will be measured in g/L at the specified time intervals.

SECONDARY OUTCOMES:
Allogeneic blood products | 12-hours post-operatively in ICU
  The volume of allogeneic blood products will be recorded.
Ventilation time | 12-hours post-operatively in ICU
  The time between intubation in OR and extubation in the ICU.
Chest tube drainage | 12-hours post-operatively in ICU
  The total volume of chest tube drainage in ICU.
Vasoactive Inotrope score | 12-hours post-operatively in ICU
  We will calculate the vasoactive inotrope score to determine if there is an increased risk of adverse outcomes.
Length of stay in ICU | Within 24 hours
  The average time of discharged from ICU.
Markers of inflammation | At 12-hours ICU
  Inflammatory mediators: tumor necrosis factor alpha (TNF-alpha), soluble receptors for advanced glycation end products (sRAGE), and high sensitivity C-reactive protein (hs CRP).
Indicators of Kidney Function | 12-hours ICU
  Serum creatinine, creatinine clearance, volume of IV fluid intake, volume of urine output, fluid balance

CONTACTS AND LOCATIONS:
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada